CLINICAL TRIAL: NCT00355134
Title: 24-month Double-blind, Randomized, Multicenter, Placebo-controlled, Parallel-group Study Comparing the Efficacy and Safety of 0.5 mg and 1.25 mg Fingolimod (FTY720) Administered Orally Once Daily Versus Placebo in Patients With Relapsing-remitting Multiple Sclerosis With Optional Extension Phase
Brief Title: Efficacy and Safety of Fingolimod (FTY720) in Patients With Relapsing-remitting Multiple Sclerosis
Acronym: FREEDOMS II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CFTY720D2309; NCT00774670 (obsolete NCT alias)
Record Dates: First submitted 2006-07-19; First posted 2006-07-21 (Estimated); Results first posted 2012-06-26 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Multiple Sclerosis
Keywords: fingolimod; FTY720; relapsing-remitting multiple sclerosis; MS; RRMS
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fingolimod 1.25 mg (Experimental): Participants received 1.25 mg fingolimod orally once a day for up to 24 months during the core phase. In the Extension phase participants continued to receive 1.25 mg fingolimod orally once a day.
  Note: Upon implementation of a protocol amendment all patients taking 1.25 mg fingolimod were switched to 0.5 mg fingolimod orally once a day.
  Interventions: Drug: Fingolimod
- Fingolimod 0.5 mg (Experimental): Participants received 0.5 mg fingolimod orally once a day for up to 24 months during the core phase. In the Extension phase participants continued to receive 0.5 mg fingolimod orally once a day.
  Interventions: Drug: Fingolimod
- Placebo (Experimental): Participants received placebo capsules orally once a day for up to 24 months during the core phase. In the Extension phase participants received either 1.25 or 0.5 mg fingolimod orally once a day.
  Note: Upon implementation of a protocol amendment all patients taking 1.25 mg fingolimod were switched to 0.5 mg fingolimod orally once a day. Upon implementation of a protocol amendment, all patients taking placebo were switched to 0.5 mg fingolimod orally once a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fingolimod — Fingolimod capsules for oral administration
  Other Names: FTY720; Gilenya®
  Arms: Fingolimod 0.5 mg; Fingolimod 1.25 mg
Drug: Placebo — Matching placebo capsules for oral administration.
  Arms: Placebo

SUMMARY:
This study assessed the safety, tolerability and efficacy of two doses of oral fingolimod compared to placebo on efficacy parameters in patients with relapsing-remitting multiple sclerosis (RRMS).

DETAILED DESCRIPTION:
This randomized, multicenter, parallel-group study consisted of 2 phases: a 24-month double-blind, randomized, multicenter, placebo-controlled, parallel-group study and an Extension phase which consisted of a dose-blinded period and an open-label period.

In the Core phase, patients were randomized to receive a fixed dose of fingolimod (0.5 mg/day), fingolimod (1.25 mg/day) or placebo for up to 24 months.

For the Extension phase, patients who were treated with fingolimod during the Core phase continued treatment at the assigned dose level, while those previously treated with placebo during the Core phase were re-randomized in a 1:1 ratio to receive one of the two doses of fingolimod (1.25 mg or 0.5 mg). All patients in the extension received blinded investigational drug: fingolimod 1.25 mg and 0.5 mg in capsules for oral administration once daily until the decision to discontinue the fingolimod 1.25 mg dose became effective and subsequently all patients were switched to open-label fingolimod 0.5 mg.

With the implementation of Amendment 11, the 1.25 mg dose was discontinued and all patients were switched to fingolimod 0.5 mg dose. With the implementation of Amendment 12, all patients treated with Placebo in the fingolimod Core phase were switched to treatment with 0.5 mg fingolimod per day. The Extension phase continued until all patients either discontinued or transferred to Study CFTY720D2399 (NCT01201356; initiated in September 2010).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between ages 18-55 with a diagnosis of multiple sclerosis
* Patients with a relapsing-remitting disease course
* Patients with expanded disability status scale (EDSS) score of 0-5.5

Exclusion Criteria:

* Patients with other chronic disease of the immune system, malignancies, acute pulmonary disease, cardiac failure, etc.
* Pregnant or nursing women

For inclusion in the extension phase patients should complete the 24 month core study with or without 24 months on study drug. If a patient discontinued study drug during the core study due to an adverse event, serious adverse event, laboratory abnormality etc. they would be excluded from the Extension Phase.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1083 (Actual)
Dates: Start 2006-06; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (112):
- United States (100):
  - University of Alabama Birmingham, Birmingham, Alabama
  - North Central Neurology Associates, PC, Cullman, Alabama
  - University of South Alabama - Dept of Neurology, Mobile, Alabama
  - Barrow Neurology Clinic, Phoenix, Arizona
  - Research and Education Institute of Alta Bates Summit Medical Center, Berkeley, California
  - University of California - Irvine, Deptarment of Neurology, Irvine, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - The Neurology Center, Oceanside, California
  - Neuro-Therapeutics, Inc., Pasadena, California
  - UC Davis Medical Center, Sacramento, California
  - Multiple Sclerosis Center at UCSF, San Francisco, California
  - University of Colorado, Denver, Colorado
  - Associated Neurologists, PC, Danbury, Connecticut
  - Associated Neurologists of Southern CT, P.C., Fairfield, Connecticut
  - Yale University - Yale Multiple Sclerosis Center, New Haven, Connecticut
  - Georgetown University Hospital - Dept of Neurology, Washington D.C., District of Columbia
  - Sunrise Clinical Research, Inc., Hollywood, Florida
  - University of Florida Health Sciences Center/Shands Jacksonville, Jacksonville, Florida
  - Neurology Associates, PA, Maitland, Florida
  - University of Miami, Department of Neurology, Miami, Florida
  - Neurological Associates, Pompano Beach, Florida
  - Roskamp Institute, Clinical Trials Division, Sarasota, Florida
  - Neurology Clinical Research, Inc, Sunrise, Florida
  - AMO Corporation, Tallahassee, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - The MS Center of Vero Beach, Vero Beach, Florida
  - MS Center of Atlanta, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Northwestern University Medical School - Dept of Neurology, Chicago, Illinois
  - Rush University Medical Center Department of Neurological Sciences, Chicago, Illinois
  - University of Chicago - Dept of Neurology, Chicago, Illinois
  - Alexian Brothers Neurosciences Research, Elk Grove Village, Illinois
  - South Suburban Neurology, Flossmoor, Illinois
  - Neurologic Associates, Ltd., Palos Heights, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Indiana University Medical Center, Indianapolis, Indiana
  - Ruan Neurology Clinical Research Center, Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Mid America Neuroscience Institute, Lenexa, Kansas
  - Kentucky Research Associates, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins MS Center, Baltimore, Maryland
  - Caritas St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Newton Wesley Hospital, Newton, Massachusetts
  - Springfield Neurology, Springfield, Massachusetts
  - UMass Memorial Medical Center, Worchester, Massachusetts
  - University of Michigan Mulitiple Sclerosis Clinic, Ann Arbor, Michigan
  - Wayne State University MS Clinic, Detroit, Michigan
  - Henry Ford Hospital, Department of Neurology, Detroit, Michigan
  - Michigan State University MS Clinic, East Lansing, Michigan
  - Michigan Medical, P.C., Grand Rapids, Michigan
  - Michigan Neurology Associates, PC, Saint Clair Shores, Michigan
  - St. Luke's Hospital - Mid-America Brain and Stroke Institute, Kansas City, Missouri
  - The MS Center for Innovation in Care, St Louis, Missouri
  - Institute for Neurosciences, Reno, Nevada
  - Multiple Sclerosis Center, Lebanon, New Hampshire
  - Gimbel Multiple Sclerosis Center at Holy Name Hospital, Teaneck, New Jersey
  - University of New Mexico Health Science Center, Albuquerque, New Mexico
  - Empire Neurology, PC, Latham, New York
  - NYU Hospital for Joint Diseases, New York, New York
  - Cornell University - NY Presbyterian Hospital, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Island Neurological Associates, PC, Plainview, New York
  - University of Rochester Medical Center, Rochester, New York
  - Alpha Neurology, Staten Island, New York
  - SUNY Stony Brook, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - UNC - Chapel Hill Neuroscience Hospital, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Neurology & Neuroscience Associates, Inc., Akron, Ohio
  - Northern Ohio Neuroscience, LLC., Bellevue, Ohio
  - NeuroCare Center, Inc, Canton, Ohio
  - River Hills Health Care, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Toledo Health Science Campus, Toledo, Ohio
  - Oak Clinic, Uniontown, Ohio
  - MS Center of Oklahoma, Mercy Neuroscience Institute, Oklahoma City, Oklahoma
  - Neurologial Associates of Tulsa, Tulsa, Oklahoma
  - Oregon Neurology, Tualatin, Oregon
  - University of Pennsylvania, Department of Neurology, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Department of Neurology, Philadelphia, Pennsylvania
  - Allegheny Neurological Associates, Pittsburgh, Pennsylvania
  - University of Pittsburgh - Dept of Neurology, Pittsburgh, Pennsylvania
  - Absher Neurology, Greenville, South Carolina
  - Mountain Empire Neurological Associates, PC, Bristol, Tennessee
  - Advanced Neurosciences Institute, Nashville, Tennessee
  - Vanderbilt Stallworth Rehabilitation Hospital, Nashville, Tennessee
  - University of Texas - Houston Medical School, Houston, Texas
  - Investigational Site - Private Practice, Lubbock, Texas
  - Integra Clinical Research, LLC, San Antonio, Texas
  - Neurology Health Care Service - Fletcher Allen Hospital, Burlington, Vermont
  - University of Virginia - Fontaine Adult Neurology, Charlottesville, Virginia
  - Virginia Mason Multiple Sclerosis Center, Seattle, Washington
  - Seattle Neuroscience Institute at Swedish Medical Center, Seattle, Washington
  - University Health Associates - West Virgina University, Morgantown, West Virginia
  - Dean Foundation, Madison, Wisconsin
  - University of Wisconsin Medical School, Madison, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
- Novartis Investigative Site, North Gosford, New South Wales, Australia
- Novartis Investigative Site, Vienna, Austria
- Canada (2):
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
- Poland (2):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Warsaw
- Romania (2):
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Târgu Mureş
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Yenisehir/Izmir
- Novartis Investigative Site, Bristol, United Kingdom

REFERENCES:
- [Derived] Wang L, Tan H, Yu J, ZhangBao J, Huang W, Chang X, Zhou L, Lu C, Xiao Y, Lu J, Zhao C, Wang M, Wu X, Wu M, Dong Q, Ngew KY, Quan C. Baseline retinal nerve fiber layer thickness as a predictor of multiple sclerosis progression: New insights from the FREEDOMS II study. Eur J Neurol. 2023 Feb;30(2):443-452. doi: 10.1111/ene.15612. Epub 2022 Nov 15. PMID 36286605
- [Derived] Fox RJ, Chan A, Zhang A, Xiao J, Levison D, Lewin JB, Edwards MR, Marantz JL. Comparative effectiveness using a matching-adjusted indirect comparison between delayed-release dimethyl fumarate and fingolimod for the treatment of multiple sclerosis. Curr Med Res Opin. 2017 Feb;33(2):175-183. doi: 10.1080/03007995.2016.1248380. Epub 2016 Nov 10. PMID 27733070
- [Derived] Derfuss T, Bergvall NK, Sfikas N, Tomic DL. Efficacy of fingolimod in patients with highly active relapsing-remitting multiple sclerosis. Curr Med Res Opin. 2015;31(9):1687-91. doi: 10.1185/03007995.2015.1067191. Epub 2015 Aug 20. PMID 26121423
- [Derived] Chinea Martinez AR, Correale J, Coyle PK, Meng X, Tenenbaum N. Efficacy and safety of fingolimod in Hispanic patients with multiple sclerosis: pooled clinical trial analyses. Adv Ther. 2014 Oct;31(10):1072-81. doi: 10.1007/s12325-014-0154-4. Epub 2014 Sep 23. PMID 25245812
- [Derived] Calabresi PA, Radue EW, Goodin D, Jeffery D, Rammohan KW, Reder AT, Vollmer T, Agius MA, Kappos L, Stites T, Li B, Cappiello L, von Rosenstiel P, Lublin FD. Safety and efficacy of fingolimod in patients with relapsing-remitting multiple sclerosis (FREEDOMS II): a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Neurol. 2014 Jun;13(6):545-56. doi: 10.1016/S1474-4422(14)70049-3. Epub 2014 Mar 28. PMID 24685276
- [Derived] Winges KM, Werner JS, Harvey DJ, Cello KE, Durbin MK, Balcer LJ, Calabresi PA, Keltner JL. Baseline retinal nerve fiber layer thickness and macular volume quantified by OCT in the North American phase 3 fingolimod trial for relapsing-remitting multiple sclerosis. J Neuroophthalmol. 2013 Dec;33(4):322-9. doi: 10.1097/WNO.0b013e31829c51f7. PMID 24051419
- See also: Fingolimod clinical trials information website — http://www.msclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were randomized to receive fingolimod 0.5 mg, 1.25 mg or placebo for up to 24 months. Upon entry into the Extension phase, patients treated with fingolimod 0.5 mg or 1.25 mg during the Core phase continued treatment at the same dose, those previously treated with placebo were re-randomized in to receive one of the two doses of fingolimod.
Groups:
- Fingolimod 1.25 mg: Participants received 1.25 mg fingolimod orally once a day for up to 24 months during the core phase. In the Extension phase participants continued to receive 1.25 mg fingolimod orally. Upon implementation of a protocol amendment, all patients taking 1.25 mg fingolimod were switched to 0.5 mg fingolimod orally once a day.
- Placebo (Core): Participants received placebo capsules orally once a day for up to 24 months during the core phase. Upon implementation of a protocol amendment, all patients taking placebo were switched to 0.5 mg fingolimod orally once a day.
- Extension: Fingolimod 1.25 mg: Participants who had received placebo in the Core phase and then received 1.25 mg fingolimod orally once a day in the Extension phase. Upon implementation of a protocol amendment, all patients taking 1.25 mg fingolimod were switched to 0.5 mg fingolimod orally once a day.
- Extension: Fingolimod 0.5 mg: Participants who had received placebo in the Core phase and then received 0.5 mg fingolimod orally once a day in the Extension phase.
Period: Core Phase
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo (Core) | Extension: Fingolimod 1.25 mg | Extension: Fingolimod 0.5 mg
Started | 370 | 358 | 355 | 0 | 0
Completed | 251 | 272 | 255 | 0 | 0
Not Completed | 119 | 86 | 100 | 0 | 0
Not completed — Withdrawal by Subject | 35 | 24 | 35 | 0 | 0
Not completed — Adverse Event | 28 | 22 | 16 | 0 | 0
Not completed — Lost to Follow-up | 17 | 13 | 21 | 0 | 0
Not completed — Abnormal laboratory value(s) | 19 | 14 | 2 | 0 | 0
Not completed — Unsatisfactory therapeutic effect | 10 | 6 | 17 | 0 | 0
Not completed — Administrative problems | 5 | 3 | 5 | 0 | 0
Not completed — Protocol Violation | 3 | 2 | 2 | 0 | 0
Not completed — Abnormal test procedure result(s) | 1 | 2 | 1 | 0 | 0
Not completed — Condition no longer requires study drug | 1 | 0 | 1 | 0 | 0
Period: Extension Phase
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo (Core) | Extension: Fingolimod 1.25 mg | Extension: Fingolimod 0.5 mg
Started | 203 | 217 | 0 | 105 | 107
Completed | 172 | 180 | 0 | 89 | 88
Not Completed | 31 | 37 | 0 | 16 | 19
Not completed — Withdrawal by Subject | 7 | 11 | 0 | 7 | 5
Not completed — Adverse Event | 13 | 9 | 0 | 3 | 5
Not completed — Lost to Follow-up | 2 | 6 | 0 | 2 | 4
Not completed — Abnormal laboratory value(s) | 4 | 2 | 0 | 2 | 2
Not completed — Administrative problems | 2 | 4 | 0 | 1 | 1
Not completed — Unsatisfactory therapeutic effect | 3 | 4 | 0 | 0 | 1
Not completed — Abnormal test procedure result(s) | 0 | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo (Core) | Extension: Fingolimod 1.25 mg | Extension: Fingolimod 0.5 mg | Total
Number analyzed (Participants) | 370 | 358 | 355 | 105 | 107 | 1295
Age Continuous [Mean (Standard Deviation); unit: years] — Demographic data for the Core phase participant population.
  years | 40.9 (8.90) | 40.6 (8.39) | 40.1 (8.42) | NA (NA) — Age demographic data presented for Core phase population only. | NA (NA) — Age demographic data presented for Core phase population only. | 40.5 (8.58)
Age Continuous [Mean (Standard Deviation); unit: years] — Demographic data for the Extension phase population. The number of participants in each treatment group in the Extension phase was 203, 217, 0, 105 and 107; Total participants 632.
  years | 40.6 (8.71) | 40.8 (7.96) | NA (NA) — Age demographic data presented for the Extension phase population only. | 39.8 (8.32) | 41.1 (8.11) | 40.6 (8.28)
Gender [Number; unit: participants] — Demographic data for the Core phase participant population.
  participants
    Female | 281 | 275 | 288 | 0 | 0 | 844
    Male | 89 | 83 | 67 | 0 | 0 | 239
Gender [Number; unit: participants] — Demographic data for the Extension phase population. The number of participants in each treatment group in the Extension phase was 203, 217, 0, 105 and 107; Total participants 632.
  participants
    Female | 148 | 160 | 0 | 88 | 85 | 481
    Male | 55 | 57 | 0 | 17 | 22 | 151

OUTCOME MEASURES:

1. Primary Outcome: Aggregate Annualized Relapse Rate (ARR) Estimate up to Month 24
Description: ARR is the average number of relapses in a year calculated by negative binomial regression as the sum of confirmed relapses of all patients in the group divided by the sum of the number of days on study of all patients in the group and multiplied by 365.25.
  A relapse was defined as the appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical demyelinating event. The abnormality must be present for at least 24 hours and occur in the absence of fever (<37.5C) or known infection. A relapse must be confirmed by the Independent Evaluating Physician (examining neurologist).
  ARR estimates were calculated from a negative binomial regression model adjusted for treatment, pooled center, number of relapses in the previous 2 years prior to enrollment, and Baseline expanded disability status scale (EDSS).
Time Frame: 24 months
Population: Full analysis set, including all patients who were randomized and took at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: relapses per year
Groups:
- Placebo: Participants received placebo capsules orally once a day for up to 24 months during the core phase. In the Extension phase participants received either 1.25 or 0.5 mg fingolimod orally once a day. Upon implementation of a protocol amendment, all patients taking 1.25 mg fingolimod were switched to 0.5 mg fingolimod orally once a day. Upon implementation of a protocol amendment, all patients taking placebo were switched to 0.5 mg fingolimod orally once a day.
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo
Number analyzed (Participants) | 370 | 358 | 355
relapses per year | 0.203 [0.165 to 0.249] | 0.208 [0.170 to 0.254] | 0.403 [0.342 to 0.475]

2. Secondary Outcome: Aggregate Annualized Relapse Rate (ARR) Estimate up to End of Study
Description: as for outcome 1
Time Frame: From Baseline until end of study (up to approximately 54 months).
Population: Core intent-to-treat (ITT) population: All patients who were randomized in the Core phase and received at least one dose of Core phase drug.
Measure: Number (95% Confidence Interval); unit: relapses per year
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo
Number analyzed (Participants) | 370 | 358 | 355
relapses per year | 0.180 [0.147 to 0.222] | 0.192 [0.157 to 0.234] | 0.363 [0.305 to 0.431]

3. Secondary Outcome: Percent Change From Baseline in Brain Volume
Description: Brain volume was measured using magnetic resonance imaging (MRI). Change from Baseline in brain volume is expressed as a percentage of the Baseline brain volume.
Time Frame: Baseline, Month 24 and end of study (up to approximately 54 months)
Population: Core intent-to-treat (ITT) population: All patients who were randomized in the Core phase and received at least one dose of Core phase drug. Patients were grouped according to the assigned treatment. "N" indicates the number of participants with data available for the specified time period.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo
Number analyzed (Participants) | 370 | 358 | 355
percent change
  Month 24 [N=247; 266; 249] | -0.595 (1.3897) | -0.858 (1.2215) | -1.279 (1.5028)
  End of study [N=178; 187; 182] | -1.130 (1.6380) | -1.266 (1.6941) | -1.694 (1.9567)

4. Secondary Outcome: Number of New or Newly Enlarged T2 Lesions
Description: Inflammatory disease activity was assessed by magnetic resonance imaging (MRI) measurement of the number of new or newly enlarged T2 lesions, by year.
Time Frame: From Baseline until Month 48
Population: Core intent-to-treat (ITT) population: All patients who were randomized in the Core phase and received at least one dose of Core phase drug. Patients were grouped according to the assigned treatment. "N" indicates the number of participants with MRI data available for the specified time period.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo
Number analyzed (Participants) | 370 | 358 | 355
lesions
  Core Phase (Month 0 to 24) [N=245; 264; 251] | 1.6 (5.41) | 2.3 (7.26) | 8.9 (13.86)
  Month 24 to 36 [N=103; 111; 102] | 0.63 (2.856) | 0.45 (1.360) | 0.63 (1.455)
  Month 36 to 48 [N=24; 15; 15] | 0.13 (0.448) | 0.07 (0.258) | 2.53 (8.741)

5. Secondary Outcome: Number of Gadolinium-enhanced T1 Lesions
Description: Inflammatory disease activity was assessed by magnetic resonance imaging (MRI) measurement of the number of gadolinium-enhanced T1 lesions.
Time Frame: Month 24 and end of study (up to approximately 54 months)
Population: Core intent-to-treat (ITT) population: All patients who were randomized in the Core phase and received at least one dose of Core phase drug. "N" indicates the number of participants with evaluable MRI data for the specified time point.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo
Number analyzed (Participants) | 370 | 358 | 355
lesions
  Core Phase (Month 24) [N=251; 269; 256] | 0.24 (2.395) | 0.37 (1.841) | 1.22 (2.967)
  End of Extension study [N=184; 194; 184] | 0.46 (2.381) | 0.09 (0.308) | 0.45 (3.618)

6. Secondary Outcome: Change From Baseline in Lesion Volume at Month 24 (Core Phase)
Description: Change from Baseline in lesion volume was measured by MRI for T2 lesions and for T1 hypointense lesions.
Time Frame: Baseline and Month 24
Population: Full analysis set for whom data were available. N=the number of patients with non-missing baseline and post-baseline values.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo
Number analyzed (Participants) | 370 | 358 | 355
mm^3
  T2 lesions [N=248, 266, 251] | -436.92 (1557.820) | -223.27 (1405.459) | 541.83 (2830.868)
  T1 hypointense lesions [N=247, 266, 248] | -99.13 (391.210) | -111.28 (530.961) | -37.68 (671.708)

7. Secondary Outcome: Percentage of Participants Free of 3-month Confirmed Disability Progression at Month 24 and End of Study
Description: Disability progression was defined using the following criteria: One point increase from baseline in patients with Baseline Expanded Disability Status Scale (EDSS) score from 0 to 5.0; or half a point increase from Baseline in patients with Baseline EDSS score of 5.5 or above. A 3-month confirmed disability progression was defined as a 3-month sustained increase from Baseline in EDSS score. The EDSS quantifies disability in multiple sclerosis in 8 functional systems; the score ranges from 0 (normal) to 10 (death due to MS). Progression curves were generated by the Kaplan-Meier method.
Time Frame: 24 months and end of study (up to approximately 54 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo
Number analyzed (Participants) | 370 | 358 | 355
percentage of participants
  At month 24 | 78.3 [73.74 to 82.87] | 74.7 [69.86 to 79.52] | 71.0 [65.94 to 76.13]
  At end of study | 66.64 [59.81 to 73.47] | 58.89 [48.98 to 68.80] | 63.51 [57.15 to 69.87]

8. Secondary Outcome: Percentage of Participants Free of 6-month Confirmed Disability Progression at Month 24 and End of Study
Description: Disability progression was defined using the following criteria: One point increase from baseline in patients with Baseline Expanded Disability Status Scale (EDSS) score from 0 to 5.0; or half a point increase from Baseline in patients with Baseline EDSS score of 5.5 or above. A 6-month confirmed disability progression was defined as a 6-month sustained increase from Baseline in EDSS score. The EDSS quantifies disability in multiple sclerosis in 8 functional systems; the score ranges from 0 (normal) to 10 (death due to MS). Progression curves were generated by the Kaplan-Meier method.
Time Frame: 24 months and end of study (up to approximately 54 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo
Number analyzed (Participants) | 370 | 358 | 355
percentage of participants
  At Month 24 | 86.9 [83.16 to 90.61] | 86.2 [82.34 to 89.97] | 82.2 [77.90 to 86.44]
  At end of study | 79.92 [74.43 to 85.41] | 74.89 [68.36 to 81.43] | 75.03 [69.59 to 80.47]

9. Secondary Outcome: Percentage of Participants Relapse-free up to Month 24
Description: Estimates of the percentage of participants relapse-free at 24 months were generated from Kaplan-Meier curves of the time to first relapse. A relapse was defined as the appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical demyelinating event. The abnormality must be present for at least 24 hours and occur in the absence of fever (<37.5C) or infection. A relapse was confirmed by an Independent Evaluating Physician.
Time Frame: 24 months
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo
Number analyzed (Participants) | 370 | 358 | 355
percentage of participants | 73.2 [68.38 to 78.01] | 71.5 [66.55 to 76.44] | 52.7 [47.20 to 58.24]

10. Secondary Outcome: Percentage of Participants Relapse-free up to End of Study
Description: Estimates of the percentage of participants relapse-free at end of study were generated from Kaplan-Meier curves of the time to first relapse. A relapse was defined as the appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical demyelinating event. The abnormality must be present for at least 24 hours and occur in the absence of fever (<37.5C) or infection. A relapse was confirmed by an Independent Evaluating Physician.
Time Frame: From Baseline until the end of study (up to approximately 54 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo
Number analyzed (Participants) | 370 | 358 | 355
percentage of participants | 63.88 [56.19 to 71.57] | 66.57 [60.86 to 72.28] | 49.12 [43.35 to 54.89]

11. Secondary Outcome: Change From Baseline in Multiple Sclerosis Functional Composite (MSFC) Z-score
Description: The Multiple Sclerosis Functional Composite (MSFC) is a multidimensional clinical outcome measure that includes quantitative tests of leg function/ambulation (Timed 25-Foot Walk), arm function (9-Hole Peg Test), and cognitive function (Paced Auditory Serial Addition Test). The overall MSFC z-score as an average of the three standardized scores derived using baseline data pooled over each treatment arm as reference population. Higher scores reflect better neurological function and a positive change from Baseline indicates improvement.
Time Frame: Baseline, Month 24 and end of study (up to approximately 54 months)
Population: Core intent-to-treat (ITT) population: All patients who were randomized in the Core phase and received at least one dose of Core phase drug. "N" indicates the number of participants with non-missing data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo
Number analyzed (Participants) | 370 | 358 | 355
units on a scale
  Month 24 [N=250; 271; 258] | -0.08 (0.916) [-6.9 to 1.3] | 0.00 (0.600) [-5.4 to 1.5] | -0.07 (0.540) [-3.6 to 1.3]
  End of Study [N=174; 187; 184] | 0.011 (0.3499) | -0.091 (0.8770) | 0.019 (0.6304)

ADVERSE EVENTS:
Time Frame: Duration of treatment was up to 24 months during the Core phase, and dependent on the length of patient participation during the Extension phase (up to approximately 54 months overall duration of treatment).
Groups:
- Core: Fingolimod 1.25 mg: Participants received 1.25 mg fingolimod orally once a day for up to 24 months during the core phase. Upon implementation of a protocol amendment, all patients taking 1.25 mg fingolimod were switched to 0.5 mg fingolimod orally once a day.
- Core: Fingolimod 0.5 mg: Participants received 0.5 mg fingolimod orally once a day for up to 24 months during the core phase.
- Core: Placebo: Participants received placebo capsules orally once a day for up to 24 months during the core phase. Upon implementation of a protocol amendment, all patients taking placebo were switched to 0.5 mg fingolimod orally once a day.
- Extension: Fingolimod 1.25 mg: Participants received 1.25 mg fingolimod orally once a day in the Extension phase. Upon implementation of a protocol amendment, all patients taking 1.25 mg fingolimod were switched to 0.5 mg fingolimod orally once a day.
- Extension: Fingolimod 0.5 mg: Participants received 0.5 mg fingolimod orally once a day in the Extension phase.
Arm/Group | Core: Fingolimod 1.25 mg | Core: Fingolimod 0.5 mg | Core: Placebo | Extension: Fingolimod 1.25 mg | Extension: Fingolimod 0.5 mg
Serious Adverse Events (participants affected / at risk) | 53/370 | 53/358 | 45/355 | 27/308 | 21/324
Other Adverse Events (participants affected / at risk) | 335/370 | 320/358 | 305/355 | 216/308 | 223/324
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core: Fingolimod 1.25 mg (N=370) | Core: Fingolimod 0.5 mg (N=358) | Core: Placebo (N=355) | Extension: Fingolimod 1.25 mg (N=308) | Extension: Fingolimod 0.5 mg (N=324)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 2 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Atrioventricular block (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 6 | 0 | 1 | 2 | 0
Cardiac flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Diabetes insipidus (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Macular oedema (Eye disorders) | 2 | 1 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Caecitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 0 | 0 | 0
Pelvic mass (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 2 | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 2 | 1 | 1 | 0
Bartholin's abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Encephalitis herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes zoster disseminated (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection fungal (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0
Vulvitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Morphoea (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 9 | 2 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Hair follicle tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Sarcoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 2 | 1 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 1 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 3 | 1 | 0 | 0
Encephalitis (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 1 | 2 | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 2 | 1 | 3 | 2 | 5
Optic neuritis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Simple partial seizures (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 2 | 1 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0
Acute psychosis (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 2 | 0 | 0
Drug dependence (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Frustration (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 3 | 0 | 0
Mania (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Paranoia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Suicidal behaviour (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1 | 1 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 3 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Cervical cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Abortion induced (Surgical and medical procedures) | 1 | 0 | 0 | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core: Fingolimod 1.25 mg (N=370) | Core: Fingolimod 0.5 mg (N=358) | Core: Placebo (N=355) | Extension: Fingolimod 1.25 mg (N=308) | Extension: Fingolimod 0.5 mg (N=324)
Lymphopenia (Blood and lymphatic system disorders) | 36 | 26 | 0 | 25 | 19
Vision blurred (Eye disorders) | 8 | 18 | 12 | 4 | 8
Abdominal pain upper (Gastrointestinal disorders) | 9 | 18 | 7 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 52 | 48 | 43 | 13 | 16
Dyspepsia (Gastrointestinal disorders) | 18 | 12 | 18 | 4 | 3
Nausea (Gastrointestinal disorders) | 57 | 63 | 54 | 13 | 14
Vomiting (Gastrointestinal disorders) | 29 | 21 | 27 | 6 | 8
Fatigue (General disorders) | 29 | 22 | 25 | 12 | 3
Pain (General disorders) | 21 | 10 | 15 | 8 | 7
Pyrexia (General disorders) | 16 | 14 | 20 | 2 | 5
Bronchitis (Infections and infestations) | 34 | 29 | 20 | 18 | 19
Influenza (Infections and infestations) | 26 | 34 | 24 | 11 | 11
Nasopharyngitis (Infections and infestations) | 88 | 84 | 85 | 50 | 52
Sinusitis (Infections and infestations) | 45 | 55 | 45 | 31 | 27
Upper respiratory tract infection (Infections and infestations) | 92 | 87 | 86 | 49 | 40
Urinary tract infection (Infections and infestations) | 45 | 47 | 54 | 23 | 24
Fall (Injury, poisoning and procedural complications) | 16 | 22 | 16 | 14 | 11
Alanine aminotransferase increased (Investigations) | 35 | 29 | 6 | 4 | 13
Gamma-glutamyltransferase increased (Investigations) | 21 | 23 | 2 | 2 | 8
Lymphocyte count decreased (Investigations) | 20 | 13 | 0 | 16 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 | 30 | 38 | 15 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 34 | 29 | 39 | 20 | 17
Neck pain (Musculoskeletal and connective tissue disorders) | 21 | 14 | 16 | 5 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 36 | 44 | 27 | 20 | 8
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 33 | 38 | 44 | 18 | 21
Dizziness (Nervous system disorders) | 53 | 38 | 43 | 10 | 11
Headache (Nervous system disorders) | 81 | 83 | 76 | 25 | 29
Migraine (Nervous system disorders) | 15 | 24 | 19 | 2 | 8
Paraesthesia (Nervous system disorders) | 14 | 19 | 18 | 5 | 5
Anxiety (Psychiatric disorders) | 18 | 18 | 17 | 5 | 5
Depression (Psychiatric disorders) | 34 | 29 | 32 | 11 | 13
Insomnia (Psychiatric disorders) | 24 | 31 | 24 | 2 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 51 | 52 | 53 | 23 | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 46 | 34 | 33 | 6 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 23 | 17 | 21 | 7 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 25 | 29 | 32 | 12 | 9
Rash (Skin and subcutaneous tissue disorders) | 21 | 22 | 24 | 14 | 12
Hypertension (Vascular disorders) | 46 | 32 | 11 | 11 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.